CLINICAL TRIAL: NCT02150889
Title: Training Effects on Fuel Metabolism
Acronym: TrainMeUpMN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1209M20741; 5R01DK098203-02 (NIH)
Record Dates: First submitted 2014-05-22; First posted 2014-05-30 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Healthy Subjects; Lean Trained Subjects; Overweight and Obesity
Keywords: insulin resistance; lipid metabolism; diabetes
MeSH Terms: conditions — Overweight; Obesity; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lean Trained (No Intervention): Metabolic control
- Obese or Overweight (Experimental): Running Program Yoga Program
  Interventions: Behavioral: Running Program; Behavioral: Yoga Program

INTERVENTIONS:
Behavioral: Running Program — 16 week supervised running program
  Arms: Obese or Overweight
Behavioral: Yoga Program — once weekly supervised yoga
  Arms: Obese or Overweight

SUMMARY:
The investigators are interested in how skeletal muscle processes fat and how this may affect insulin resistance. This is an important question since insulin resistance predates and predicts type 2 diabetes. The investigators are especially interested in learning about the effects of weight and training on insulin resistance. The investigators will study people before and after supervised aerobic or yoga training to identify differences in resting fat and sugar metabolism which may lead to differences in insulin resistance. The investigators will test these differences using stable isotopes, and the use of these stable isotopes is experimental.

Overweight/Obese Group: Eight visits will be required at the University of Minnesota Clinical Research Unit. Four visits will be done before training (screen and 3 pre-training visits), 1 visit during the training, and 3 post-training visits will be done. In between, the training will take about 16 weeks and will be a supervised treadmill program.

Lean/Trained Group: Four visits will be required at the University of Minnesota Clinical Research Unit (screen and 3 study visits).

DETAILED DESCRIPTION:
Insulin resistance plays a critical role in the development of type 2 diabetes (T2DM), with skeletal muscle the largest site of insulin resistance in the human body. In sedentary humans, insulin resistance correlates with levels of intramyocellular lipid (IMCL) and lipid metabolites that adversely affect skeletal muscle glucose metabolism. However, even modest endurance training has been shown to reduce insulin resistance while increasing skeletal muscle IMCL. Moreover, lean endurance trained participants have IMCL levels comparable to those of patients with T2DM, yet have significantly lower insulin resistance. These findings suggest that the physiological changes caused by training protect against lipid induced insulin resistance and that this protection is present even at rest, however our preliminary data suggest that training facilitates utilization of readily available fuel, with lipid preferentially used over glucose when available. We will test the overarching hypothesis that training increases resting skeletal muscle lipid metabolism, as measured by markers of IMCL lipolysis, accumulation of fatty acid metabolites and mitochondrial utilization of fatty acids.

Research reported in this publication was supported by the National Center for Advancing Translational Sciences of the National Institutes of Health Award Number UL1-TR002494. The content is solely the responsibility of the authors and does not necessarily represent the official views of the National Institutes of Health.

ELIGIBILITY:
Inclusion Criteria:

All subjects

1. Subjects 18 to 40 years of age.
2. Subjects are capable of giving informed consent

Overweight or obese

1. Insulin resistant based on screening oral glucose tolerance testing.
2. BMI 25 to 40 kg/m2 inclusive
3. Stable weight for at least 3 months (± 5 lbs.)
4. Sedentary status (self-report < 30 minutes/week regular exercise).

Lean, physically active

1. physically active subjects defined as 3-5 aerobic exercise sessions/week
2. matched to age and gender
3. generally healthy with normal fasting glucose levels (glucose ≤100 mg/dL).

Exclusion Criteria:

All subjects

1. Subjects 18 to 40 years of age.
2. Subjects are capable of giving informed consent

Overweight or obese

1. Insulin resistant based on screening oral glucose tolerance testing.
2. BMI 25 to 40 kg/m2 inclusive
3. Stable weight for at least 3 months (± 5 lbs.)
4. Sedentary status (self-report < 30 minutes/week regular exercise).

Lean, physically active

1. physically active subjects defined as 3-5 aerobic exercise sessions/week
2. matched to age and gender
3. generally healthy with normal fasting glucose levels (glucose ≤100 mg/dL).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in insulin sensitivity between groups | Before and after exercise program (exercise program will take 16 weeks, expected average for evaluation will be 20 weeks)
  Will use HOMA-IR and hyperinsulinemia-euglycemic clamp

SECONDARY OUTCOMES:
Differences in fitness level between groups | before and after exercise program (exercise program will take 16 weeks, expected average for evaluation will be 20 weeks)
  we will measure fitness level by treadmill based VO2 max testing.

OTHER OUTCOMES:
Differences in body composition between groups | before and after exercise program ((exercise program will take 16 weeks, expected average for evaluation will be 20 weeks)
  we will measure body composition by iDEXA to look at changes and total fat, visceral fat, and subcutaneously pre-and post exercise. This will be a noninvasive x-ray based measurement (x-ray exposure is extremely low and is equivalent to 1 day of natural radiation in Minnesota)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S. Chow, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Nelson AB, Chow LS, Stagg DB, Gillingham JR, Evans MD, Pan M, Hughey CC, Myers CL, Han X, Crawford PA, Puchalska P. Acute aerobic exercise reveals that FAHFAs distinguish the metabolomes of overweight and normal-weight runners. JCI Insight. 2022 Apr 8;7(7):e158037. doi: 10.1172/jci.insight.158037. PMID 35192550
- [Derived] Bantle AE, Bosch TA, Dengel DR, Wang Q, Mashek DG, Chow LS. DXA-Determined Regional Adiposity Relates to Insulin Resistance in a Young Adult Population with Overweight andObesity. J Clin Densitom. 2019 Apr-Jun;22(2):287-292. doi: 10.1016/j.jocd.2018.06.001. Epub 2018 Jun 7. PMID 30064815